CLINICAL TRIAL: NCT04093934
Title: Developing a Sustainable Organizational Structure to Integrate Psychosocial Stimulation Programme Into Primary Health Care Services in Bangladesh [Bangladesh Undertaking Child Development and Health-system Integration (BUDHI) Project]
Brief Title: Strengthening Bangladeshi Babies Brains (SBBB)
Acronym: BUDHI/SBBB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bangor University (Other); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-19040
Record Dates: First submitted 2019-08-18; First posted 2019-09-18 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-01

CONDITIONS: Child Development
Keywords: Early childhood development; Psychosociaal stimulation; Bayley test; Bangladesh; Undernutrition; Stepped wedge design; Cluster randomized controlled trial
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Support

STUDY DESIGN:
Intervention Model Description: 'stepped wedge design'
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Children in the intervention arm will receive sessions of psychosocial stimulation every two weeks at the community clinics for one year. The intervention includes songs, games, book and toy activities for undernourished children and nutritional and developmental messages for their mothers.
  Interventions: Behavioral: Psychosocial stimulation
- Wait-listed control (No Intervention): The wait-listed controls will be only tested at baseline and after a year. Following completion of the 2nd test, they will be included in the study and receive the same intervention provided to children in the experimental arm.

INTERVENTIONS:
Behavioral: Psychosocial stimulation — Children will receive fortnightly sessions of psychosocial stimulation and nutritional support for one year during the study period.
  Other Names: Nutritional support
  Arms: Intervention

SUMMARY:
This study aims to establish a sustainable programme whereby early childhood development activities are integrated into the routine activities of community clinics in rural Bangladesh for undernourished children by developing a cascade of training at national, district, Upazila (sub-district), and union level to train clinic staff.

DETAILED DESCRIPTION:
Background (brief):

1. Burden: Approximately 250 million children under 5 years of age in developing countries do not reach their full potential due to poverty, malnutrition and lack of a stimulating environment. It is estimated that in Bangladesh 44% of the population live below the international poverty line, and 36% of children under 5 years are stunted. Bangladeshi children showed a significant cognitive deficit as early as 7 months of age compared to more affluent children and the deficit grew bigger as children reached 5 years of age.
2. Knowledge gap: Several studies in developing countries have shown benefits of early childhood interventions to development of under-5 children. The curriculum of early childhood intervention 'Reach up' has been adapted for Bangladesh and used in 6 trials in Bangladesh. All the projects found consistent significant benefits on the developmental outcomes of children. Two recent trials were conducted in community clinics (CCs), integrating early childhood development (ECD) activities with Govt primary health service and there is a need to determine if the intervention can be taken to scale.
3. Relevance:

Bangladesh Govt acknowledges the need for improving children's development and has agreed to collaborate and implement ECD activities at large scale in addition to funding it.

Hypothesis (if any): We hypothesize that it is feasible to train GoB staff at District, Upazila (Sub-district), Union and CC levels and integrate ECD activities in CCs in Bangladesh and thereby improve undernourished children's development after a year of intervention.

Objectives:

1. To establish an organizational structure for the programme to be sustainable
2. To establish a mechanism for sustainability at national, district and Upazila levels: including training, supervision, monitoring and reporting
3. To assess the impact on maternal knowledge and depressive symptoms, stimulation in the home and child growth, cognition and language in a subsample

Methods: Undernourished children aged 6-24 months will be identified using mid-arm upper circumference (MUAC) by Govt. Health staff in 12 Upazilas of Sylhet and 11 Upazilas of Chittagong Divisions. We target to include 554 Community clinics in the programme and train approx. 1600 CC staff to deliver the parenting session. We will evaluate a subsample of the children through a 'stepped wedge design' to assess the effects of intervention using a cluster randomized controlled trial.

Outcome measures/variables: The main outcomes are coverage, compliance and fidelity of the programme. In addition, children's cognitive and language development and behaviour will be assessed in a sub-sample.

ELIGIBILITY:
Inclusion Criteria:

* Moderately and severely malnourished children
* Aged 6-24 mo
* Both sexes
* Mid-upper arm circumference (MUAC)<12.5 cm
* Parents agree to participate in the programme.

Exclusion Criteria:

* Children with MUAC≥12.5 cm
* Those whose parents do not consent to participate
* Children with disability, multiple births or any congenital abnormality will be included in the intervention but excluded from the evaluation sample

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Through study completion, an average of 1 year
  Cognitive Composite scores on Bayley Scales of Infant and Toddler Development-III test, measuring children's cognition aged 1-42 months, ranging from 55 to 145. Higher values represent better outcome.
Language development | Through study completion, an average of 1 year
  Language Composite scores on Bayley Scales of Infant and Toddler Development-III test, measuring children's language aged 1-42 months, ranging from 47 to 153. Higher values represent better outcome.

SECONDARY OUTCOMES:
Response to examiner | Through study completion, an average of 1 year
  Wolke's Behaviour ratings measuring response to examiner of children aged 1-42 months ranging from 1-9. Higher values represent better outcome.
Emotional Tone | Through study completion, an average of 1 year
  Wolke's Behaviour ratings measuring emotional tone of children aged 1-42 months ranging from 1-9. Higher values represent better outcome.
Cooperation with test procedure | Through study completion, an average of 1 year
  Wolke's Behaviour ratings measuring cooperativeness of children aged 1-42 months ranging from 1-9. Higher values represent better outcome.
Vocalization | Through study completion, an average of 1 year
  Wolke's Behaviour ratings measuring vocalization of children aged 1-42 months ranging from 1-9. Higher values represent better outcome.
Quality of home stimulation | Through study completion, an average of 1 year
  Family Care Indicators (FCI), measuring play activities (ranging from 0-15), play materials (ranging from 0-7), books (ranging from 0-10), and magazines (ranging from 0-10), available to child at home. The sub-scales of play activities, play materials, books and magazines will be summed to make a total FCI score, ranging from 0-42. Higher values represent better outcome.
Anthropometry | Through study completion, an average of 1 year
  WHO standards for measuring weight in kilograms, length/height and head circumference in centimeters. These measures will be converted to Z scores for head-circumference-for-age, weight-for-age, length/height-for-age and weight-for-length/height. Values between - to +1 Z scores represent normal values and increment up to +3 Z score represent improvement. But, values more than +3 Z score are not normal.
Maternal knowledge of child rearing | Through study completion, an average of 1 year
  Pre-designed and previously used questionnaire measuring maternal knowledge of child development, ranging from 0-50. Higher values represent better outcome.
Maternal depressive symptoms | Through study completion, an average of 1 year
  Family Care Indicators measuring 6 depressive symptoms of mothers in days for the last 7 days, ranging from 0-42. Lower values represent better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jena D Hamadani, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
The data will not be shared with other researchers in its present form, however, de-identified data may be shared with other researchers if they come up with any novel idea for new analysis.

REFERENCES:
- [Derived] Tipu SMMU, Hossain SJ, Arifeen SE, Mehrin SF, Salveen NE, Kawsir M, Bhuiyan MSA, Shiraji S, Hasan MI, Tofail F, Hamadani JD. A sustainable organizational structure to integrate psycho-social stimulation programme into primary health care services in Bangladesh: protocol for a pragmatic cluster randomized controlled trial on scaling up early childhood development activities. BMC Psychol. 2025 May 19;13(1):525. doi: 10.1186/s40359-025-02795-w. PMID 40390132